CLINICAL TRIAL: NCT07303738
Title: The Use of High Bile-Binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations: A Novel Intervention for Children at Risk for Aspiration-Associated Complications (Aim 1)
Brief Title: The Use of High Bile-binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations (Aim 1)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Director, Aerodigestive Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00049734 Aim 1
Expanded Access: Available
Record Dates: First submitted 2025-03-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-03

CONDITIONS: Feeding Difficulties; Aspiration; Gastrostomy
Keywords: blenderized; bile acid; gastrostomy; aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- amino acid-based formula (e.g., elecare, neocate) (Active Comparator)
  Interventions: Drug: amino acid based formula (e.g. Elecare Jr)
- low bile acid binding blenderized diet (e.g., real food blends) (Active Comparator)
  Interventions: Drug: low bile acid binding blenderized diet (e.g. Kate Farms)
- high bile acid binding blenderized diet (proprietary) (Experimental)
  Interventions: Drug: high bile acid binding blenderized diet

INTERVENTIONS:
Drug: amino acid based formula (e.g. Elecare Jr) — We will administer one bolus of an amino acid based formula
  Arms: amino acid-based formula (e.g., elecare, neocate)
Drug: low bile acid binding blenderized diet (e.g. Kate Farms) — We will administer one bolus of a low bile acid binding blenderized diet
  Arms: low bile acid binding blenderized diet (e.g., real food blends)
Drug: high bile acid binding blenderized diet — We will administer one bolus of a high bile acid binding blenderized diet
  Arms: high bile acid binding blenderized diet (proprietary)

SUMMARY:
We will perform an acute physiology study comparing three different diets-an amino acid-based formula, a low bile acid-binding blenderized diet, or a high bile acid-binding blenderized diet administered through gastrostomy tube. We will determine the differences in gastric and salivary bile acid concentrations between participants over the 4 hour post-prandial timeframe.

Participants who regularly receive an amino acid-based formula will receive an amino acid-based formula during the study and participants who regularly receive a blenderized feed will receive a blenderized feed during the study. Only participants who regularly receive blenderized feeds will be randomized to receive either the high or low bile acid binding blenderized feed.

ELIGIBILITY:
Inclusion Criteria:

* receive at least 80% of their nutritional needs by gastrostomy
* receive either an amino acid-based formula, an International Dysphagia Diet Standardization Initiative level 4 commercial blend, or a home blend
* can receive bolus feeds of 240 cc within 30 minutes or less

Exclusion Criteria:

* have received a fundoplication
* receive post-pyloric feeds
* require medication/flush administration during the four-hour study period
* are allergic to any component of the study diets.

To participate in this study, if patients are taking acid suppression or motility medications (e.g., erythromycin, azithromycin, prucalopride), they will need to stop these at least 72 hours prior to participation in this aim.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Gastric bile acid concentration | 4 hours
  Mean difference in gastric bile acid concentrations between start of feed and four hours following feed

SECONDARY OUTCOMES:
Gastric bile acid concentration | 1, 2 and 3 hours
  Differences in gastric bile acid concentrations from start of feed to 1, 2 and 3 hours after feed between groups
Correlations between gastric bile acid and gastroesophageal reflux Likert scale | Baseline to 1, 2, 3 and 4 hours post-prandial
  Correlations between the postprandial changes in gastric bile acid concentrations and gastroesophageal reflux Likert scores
Correlation of symptom scores with gastric and salivary bile acid concentration | baseline
  comparison of PedsGIQL scores, GERD Likert scores, and PC-QoL scores with baseline gastric and salivary bile acid concentrations
Correlation of gastric and salivary bile acid concentrations | 0, 1, 2, 3 and 4 hours post-prandial
  correlations between gastric and salivary bile acid concentrations at each time point
correlations between C13 excretion rates and gastric and salivary bile acid concentrations | Baseline to 1, 2, 3 and 4 hours post-prandial
  correlations between C13 excretion rates and gastric and salivary bile acid concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No